CLINICAL TRIAL: NCT03855332
Title: Oxford Haemodynamic Adaptation to Reduce Pulsatility: Randomised, Placebo-controlled, Double-blind Crossover Trial of Effects of Sildenafil on Cerebral Arterial Pulsatility in Patients With Cryptogenic or Lacunar Stroke and Small Vessel Disease
Brief Title: Oxford Haemodynamic Adaptation to Reduce Pulsatility Trial
Acronym: OxHARP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13891; 206589/Z/17/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2019-02-21; First posted 2019-02-26 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2022-05

CONDITIONS: Small Vessel Cerebrovascular Disease
MeSH Terms: conditions — Cerebral Small Vessel Diseases | interventions — Sildenafil Citrate; Cilostazol

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, placebo and active controlled, crossover design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): All participants will undergo three phases in random order:
  The placebo phase will include overencapsulated placebo, matched to overencapsulated active agents, 2 tablets 3 times daily
  Interventions: Drug: Placebo
- Sildenafil (Experimental): 25mg three times daily, overencapsulated tablet, increased after 1 week to 50mg three times daily
  Interventions: Drug: Sildenafil
- Cilostazol (Active Comparator): 50mg bd, overencapsulated tablet (with midday placebo), increased after 1 week to 100mg bd (with midday placebo)
  Interventions: Drug: Cilostazol

INTERVENTIONS:
Drug: Sildenafil — See above
  Arms: Sildenafil
Drug: Cilostazol — See above
  Arms: Cilostazol
Drug: Placebo — Overencapsulated placebo
  Arms: Placebo

SUMMARY:
Chronic damage to small blood vessels deep in the brain is seen in half of patients over the age of 60 and almost all patients over the age of 80, and is responsible for up to a third of strokes and almost half of patients with dementia. However, there is limited evidence for how small vessel disease develops and no specific treatment. One potential explanation is that greater pulsations in blood pressure are transmitted to the brain through stiff blood vessels, resulting in increased pressure hitting the brain each time the heart beats and reduced blood flow between heart beats.

Sildenafil is used to open up blood vessels (a vasodilator) in patients with erectile difficulties or poor blood supply to the lungs. This trial will test sildenafil (50mg, thrice daily) against placebo and a similar drug (cilostazol 100mg, twice daily) in 75 patients with previous stroke or mini-stroke and small vessel disease, given in random order to every participant for 3 weeks each. It will primarily assess changes in pulsations of blood flow to the brain on each tablet, measured with an ultrasound scanner (transcranial ultrasound). To understand why any changes occur, we will also measure the stiffness of arteries, the blood pressure at the heart and how much blood vessels in the brain open up when participants breathe air with added carbon dioxide (6%), using ultrasound in all participants and on MRI brain scans in 30 patients.

This study will test whether a vasodilator used in other conditions with a good safety profile can reduce pulsations in blood flow to the brain, to assess whether it is a good candidate drug to reduce the progression of small vessel disease in future clinical trials. This would be the first effective treatment for a condition associated with a very high burden of disability.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Can record MCA waveform on at least one side ('useable TCD window')
* Non-disabling, ischaemic stroke or TIA, >1 month prior to randomisation, of either cryptogenic or lacunar aetiology, confirmed clinically or on brain imaging
* White matter hyperintensities on MRI (Fazekas scale) or CT (Blennow scale) consistent with cerebral small vessel disease
* Age below 60 MRI Fazekas score 1 to 3 (max 2 points in periventricular or deep score) or CT Blennow score 1 to 3 (max 2 points in periventricular or deep score)
* Age above 60 MRI Fazekas score 1 to 4 (max 2 points in periventricular or deep score) or CT Blennow score 1 to 4 (max 2 points in periventricular or deep score)

Exclusion Criteria:

* Pregnant or breastfeeding women, women of childbearing age not taking contraception.
* Other major neurological or psychiatric conditions affecting the brain and interfering with the study design (e.g. multiple sclerosis)
* Other causes of stroke such as

  * ≥50% luminal stenosis (NASCET) in large arteries supplying the infarct area
  * major-risk cardioembolic source of embolism (permanent or paroxysmal atrial fibrillation, sustained atrial flutter, intracardiac thrombus, prosthetic cardiac valve, atrial myxoma or other cardiac tumours, mitral stenosis, recent (<4 weeks) myocardial infarction, left ventricular ejection fraction less than 30%, valvular vegetations, or infective endocarditis)
  * other specific causes of stroke (e.g. arteritis, dissection, drug misuse)
* Large vessel occlusion on MRA or CTA (carotid, basilar or MCA)
* Modified Rankin Score >3
* Unable to swallow
* Renal impairment (eGFR <35ml/min)
* Significant biochemical abnormalities (sodium <130, K+ <2.5 or >5.5, LFTs >3 x upper limit of normal range)
* Life expectancy <2 years
* Contraindication to active agents

  * Concurrent use of alphablocker
  * Regular use of nitrate (ISMN, GTN, other)
  * Heart failure (NYHA 2-4)
  * Severe aortic stenosis
  * Bilateral renal artery stenosis
  * Uncontrolled arrhythmias
  * Previous priapism
  * Anatomical deformation of the penis
  * Recent myocardial infarction (within 6 months)
  * Unstable angina
  * History of non-arteritic ischaemic optic neuropathy
  * Hypotension: BP <90/60
  * Haemodynamically significant aortic / mitral valve disease
  * Sickle cell disease, myeloma, leukaemia
  * Uncontrolled hypertension (BP >180/110 despite treatment with 3 antihypertensives)
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study or the participant's ability to participate in the study.
* Participants who have participated in another research study involving an investigational product in the past 12 weeks.
* Use of an anticoagulant (warfarin, dabigatran, rivaroxaban etc) or more than one antiplatelet drug.
* Predisposition to intracerebral haemorrhage (previous ICH, likely cerebral amyloid angiopathy) or intraocular haemorrhage (uncontrolled diabetic retinopathy or neovascularisation)
* Allergy to constituents of medications or components of placebo / overencapsulation
* Use of CYP inducers that interact with study medications (ketoconazole, erythromycin).

Exclusion criteria specific for MRI substudy

* Not able to transfer to MRI scanner
* Active respiratory illness (such as moderate to severe asthma or COPD) such that they are unable to tolerate MRI or unable to lie flat
* Claustrophobia
* Contraindication to MRI scan (pacemaker, aneurysm clip etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Middle cerebral arterial pulsatility index | 3 weeks
  Difference in Gosling's pulsatility index after three weeks treatment with sildenafil versus placebo, in 75 patients

SECONDARY OUTCOMES:
Percentage increase in MCA velocity on 6% CO2 vs medical air | 3 weeks
  1. Difference in cerebrovascular reactivity after 3 weeks of treatment with sildenafil versus placebo in 75 patients: cereborovascular reactivity calculated by the percentage increase in mean MCA velocity whilst breathing 6% CO2 compared to breathing medical air.
  2. Non-inferiority of 3 weeks of treatment with cilostazol 100mg bd compared to sildenafil 50mg tds for difference in Gosling's pulsatility index and cerebrovascular reactivity to 6% CO2.

OTHER OUTCOMES:
Reactivity of BOLD signal on MRI to 6% CO2 challenge | 3 weeks
  Difference in cerebrovascular reactivity after 3 weeks of treatment with sildenafil versus placebo in 30 patients: cerebrovascular reactivity calculated by the percentage increase in BOLD signal on MRI whilst breathing 6% CO2 compared to breathing medical air.

CONTACTS AND LOCATIONS:
Overall Officials: Dr A Webb, DPhil, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, Oxon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
This will be determined on specific request

REFERENCES:
- [Derived] Webb AJ, Feakins K, Lawson A, Stewart C, Thomas J, Llwyd O. White matter hyperintensities are independently associated with systemic vascular aging and cerebrovascular dysfunction. Int J Stroke. 2025 Jun;20(5):581-589. doi: 10.1177/17474930241306987. Epub 2025 Jan 3. PMID 39614707
- [Derived] Webb AJS, Birks JS, Feakins KA, Lawson A, Dawson J, Rothman AMK, Werring DJ, Llwyd O, Stewart CR, Thomas J. Cerebrovascular Effects of Sildenafil in Small Vessel Disease: The OxHARP Trial. Circ Res. 2024 Jul 5;135(2):320-331. doi: 10.1161/CIRCRESAHA.124.324327. Epub 2024 Jun 4. PMID 38832504
- [Derived] Webb A, Werring D, Dawson J, Rothman A, Lawson A, Wartolowska K. Design of a randomised, double-blind, crossover, placebo-controlled trial of effects of sildenafil on cerebrovascular function in small vessel disease: Oxford haemodynamic adaptation to reduce pulsatility trial (OxHARP). Eur Stroke J. 2021 Sep;6(3):283-290. doi: 10.1177/23969873211026698. Epub 2021 Jun 23. PMID 34746425

DOCUMENTS (2):
  • Study Protocol (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT03855332/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT03855332/SAP_001.pdf